CLINICAL TRIAL: NCT06097429
Title: Evaluation of Platelet Aggregation in COVID-19 Patients
Brief Title: Platelet Aggregation in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MS.21.07.1596
Record Dates: First submitted 2023-10-20; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: platelet aggregation; COVID-19; ADP; light-transmission aggregometry
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection; Platelet Aggregation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: COVID-19 confirmed cases with positive PCR test in the first week of diagnosis
  Interventions: Diagnostic Test: blood sample for platelet aggregation
- control group: healthy volunteers, persons with no history nor symptoms suggestive of COVID-19 with negative COVID -19 PCR test and no CT Chest changes suggestive of COVID-19 infection.
  Interventions: Diagnostic Test: blood sample for platelet aggregation

INTERVENTIONS:
Diagnostic Test: blood sample for platelet aggregation — evaluate platelet aggregation using light-transmission aggregometry and adenosine diphosphate (ADP)

SUMMARY:
Context: Hypercoagulable state associated with COVID-19 is one of the pathologic events that noticed in different waves of COVID-19 pandemics and leads to serious consequences in mortality and morbidity Aim: To evaluate platelet aggregation using light-transmission aggregometry and adenosine diphosphate (ADP) as an agonist in COVID-19 patients.

Settings and design: This was prospective cross-sectional study. Patients and methods: Seventy-five individuals were enrolled in this study and divided into two groups, 50 patients with PCR-positive COVID-19 as study group and 25 apparently healthy individual as a control group. All individuals were subjected to full clinical evaluation, CT-chest, laboratory investigations: CBC, INR, LDH, CRP, serum ferritin and platelet aggregation evaluation using light-transmission aggregometry and adenosine diphosphate (ADP) as an agonist

DETAILED DESCRIPTION:
This observational, case control study included 50 adult patients with positive COVID-19 PCR test recruited from isolation department of Mansoura university hospital from July 2021 to May 2022 as a study group, and control group included 25 healthy persons with no history nor symptoms of COVID -19 and negative PCR test, matched with the study group regarding the demographic variables and comorbidities.

The protocol of this study was approved by the Institutional Research Board of Faculty of Medicine, Mansoura University (code no: MS.21.07.1596) and written informed consents were obtained from all patients to be enrolled in this study.

The aim of this study was to evaluate platelet aggregation using light-transmission aggregometry and adenosine diphosphate (ADP) as an agonist in COVID-19 patients, in comparison to that in healthy controls.

Patients:

Inclusion criteria:

Age ≥ 18 years old.

Study group: COVID-19 confirmed cases with positive PCR test in the first week of diagnosis with COVID-19 CT changes with any severity grade according to WHO, (2020) as:

Mild cases: mild clinical symptoms and no imaging findings of pneumonia. Moderate cases: fever, respiratory symptoms and radiological abnormalities of COVID-19.

Severe cases: meet any of the following; SpO2 < 93%, PaO2 /FiO2 < 300, respiratory rate equal or more than 30 breaths/min, or lung infiltration more than 50% including GGO or consolidation .

Critically ill cases: respiratory failure, need for invasive MV, septic shock, and/or multiorgan dysfunction.

Exclusion criteria:

The following patients were excluded:

Patients with thrombocytopenia and thrombocytosis defined as platelet count less than 100,000/ µL, count more than 450,000 / µL respectively Patients with hematocrit abnormalities as less than 34% or greater than 55% Patients with disseminated intravascular coagulation (DIC) Active malignancy Liver disease as such chronic hepatitis, cirrhosis or liver cell failure. Any hematological disorders as hemophilia or thalassemia. Patients on invasive mechanical ventilation as endotracheal intubation and mechanical ventilation itself are factors for having a higher mean platelet volume (MPV) which means that platelets are larger than average which are more adhesive and likely to aggregate in vitro. Patients receiving aspirin, non-steroidal anti-inflammatory drugs, antiplatelet drugs or any other medications that can influence platelet function (14 days prior to blood sample collection)

Control group: healthy volunteers, persons with no history nor symptoms suggestive of COVID-19 with negative COVID -19 PCR test and no CT Chest changes suggestive of COVID-19 infection. They were also matched with the study group in demographic variables and comorbidities. Methods:

All patients were subjected to the following:

1. Full history taking with stress on: Demographic data (age and sex), smoking history and co-morbid diseases as chronic obstructive pulmonary disease, hypertension, diabetes mellitus, ischemic heart disease, bronchial asthma, cerebral stroke, and malignancy. Symptoms suggestive of COVID-19 as dyspnea, cough, expectorations, hemoptysis, fever, bone aches, sore throat, loss of taste, anosmia, diarrhea and headache.
2. General and local chest examination.
3. Laboratory investigations as:

   1. Complete blood count (CBC)
   2. Liver function tests (ALT, AST, and serum albumin)
   3. Serum creatinine • International normalized ratio (INR).
   4. Inflammatory markers as (lactate dehydrogenase (LDH), C- reactive protein (CRP), D-dimer and serum ferritin)
4. Radiological assessment (CT chest):

   i. Description either consolidation or ground glass opacity according to Hansell et al. (2008).

   ii. CT severity score was assessed according to Bernheim et al. (2020) with each of the five lung lobes assessed and scored for the degree of involvement and classified as: score 0, no involvement (0% affected); 1, minimal (1%-25%); 2, mild (26%-50%); 3, moderate (51%-75%); and 4, severe (76%-100%). A total severity score was obtained by summing the five lobe scores, with a range between 0 and 20. A score of 1-5 was graded as "minimal," 6-10 as "mild," 11-15 as "moderate," and 16-20 as "severe."
5. Platelet aggregation work:

   1. Reagent used: Adenosine diphosphate (ADP) was used in this study as an agonist to enhance and evaluate platelet aggregation. It is a lyophilized preparation of adenosine-5'-diphosphate. The working concentration of the reconstituted reagent is 200 µM.
   2. Device of aggregation: a platelet lighttransmission aggregometer (PAP-8E brand aggregometer). It is manufactured by Bio/Data Corporation in USA, it has programmable electronic pipette with charging stand, 8 test channels and computer with monitor.
   3. Test procedure was done according to Hvas and Favaloro (2017)
6. Outcomes measures:

   1. Developing new thromboembolic event as arterial or venous thrombosis, such as acute myocardial infarction (AMI), cerebral stroke, and pulmonary thromboembolism during hospitalization and specifying the type of this event.
   2. Need to invasive mechanical ventilation (MV).
   3. Length of hospital stay (days) including more or less and equal 7 days.
   4. Mortality rate.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old.

Exclusion Criteria:

* • Patients with thrombocytopenia and thrombocytosis defined as platelet count less than 100,000/ µL, count more than 450,000 / µL respectively

  * Patients with hematocrit abnormalities as less than 34% or greater than 55%
  * Patients with disseminated intravascular coagulation (DIC)
  * Active malignancy
  * Liver disease as such chronic hepatitis, cirrhosis or liver cell failure.
  * Any hematological disorders as hemophilia or thalassemia.
  * Patients on invasive mechanical ventilation as endotracheal intubation and mechanical ventilation itself are factors for having a higher mean platelet volume (MPV) which means that platelets are larger than average which are more adhesive and likely to aggregate in vitro. Patients receiving aspirin, non-steroidal anti-inflammatory drugs, antiplatelet drugs or any other medications that can influence platelet function (14 days prior to blood sample collection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study group: COVID-19 confirmed cases with positive PCR test in the first week of diagnosis with COVID-19 CT changes with any severity grade according to WHO, (2020)
  Control group: healthy volunteers, persons with no history nor symptoms suggestive of COVID-19 with negative COVID -19 PCR test and no CT Chest changes suggestive of COVID-19 infection. They were also matched with the study group in demographic variables and comorbidities.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Mortality rate. | day 0 to day 30
  recording from any mortality from the study and the control group

SECONDARY OUTCOMES:
Developing new thromboembolic event as arterial or venous thrombosis | day 0 to day 30
  acute myocardial infarction (AMI), cerebral stroke, and pulmonary thromboembolism during hospitalization and specifying the type of this event
Need to invasive mechanical ventilation (MV) | day 0 to day 30
  number of cases deteriorating and managed by invasive mechanical ventilation
Length of hospital stay (days) | day 0 to day 30
  more or less and equal 7 days

CONTACTS AND LOCATIONS:
Overall Officials: rehab Ah elmorsey, MD, Study Chair — Mansoura University, chest medicine departmenr
Locations (1):
- Faculty of Medicine, Al Mansurah, Egypt